CLINICAL TRIAL: NCT00004728
Title: Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) Study
Brief Title: Aspirin Or Warfarin To Prevent Stroke
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: R01NS036643 (NIH)
Record Dates: First submitted 2000-02-25; First posted 2000-02-28 (Estimated); Last update posted 2006-06-06 (Estimated); Status verified 2006-06

CONDITIONS: Stroke; Cerebral Infarction; Atherosclerosis; Constriction, Pathologic
Keywords: stroke; cerebral infarction; warfarin; coumadin; aspirin; ASA; acetysalicylic acid; atherosclerosis; stenosis; intracranial; artery; arteries; transient ischemic attack; TIA; minorities
MeSH Terms: conditions — Stroke; Cerebral Infarction; Atherosclerosis; Constriction, Pathologic; Ischemic Attack, Transient | interventions — Warfarin; Aspirin

INTERVENTIONS:
Drug: Warfarin
Drug: Aspirin

SUMMARY:
The purpose of this study is to determine whether aspirin or warfarin is more effective in preventing stroke in patients with intracranial stenosis.

DETAILED DESCRIPTION:
Prevention of stroke in patients with narrowing of one of the arteries in the brain typically consists of using medications to prevent blood clots from forming. Currently, the best medication to use in this situation is unknown. The purpose of this study is to compare the effectiveness of two different medications, warfarin or aspirin, for the prevention of stroke due to narrowing of one of the large arteries in the brain. Patients must have experienced a recent transient ischemic attack (TIA) or mild stroke. Stroke of this type is thought to occur more often in minorities.

ELIGIBILITY:
Inclusion Criteria:

* TIA or non-severe stroke within 90 days prior to randomization (including day 90)
* Modified Rankin score of < 3
* High grade stenosis (50 to 99 percent) of a major intracranial artery (carotid artery, MCA stem (M1), vertebral artery,and basilar artery) documented by conventional angiography within 90 days prior to randomization (including day 90)
* TIA or stroke is attributed to high grade intracranial stenosis
* Age > 40 years
* Patient is able to follow an outpatient protocol(requiring monthly blood tests and clinic visits every four months for the duration of the study) and is available by telephone
* Patient understands the purpose and requirements of the study, can make him/herself understood, and has provided informed consent

Exclusion Criteria:

* Extracranial carotid stenosis (> 50 percent) ipsilateral to stenosis of the intracranial carotid artery or MCA (ie.tandem stenoses, either of which could have caused patient's symptoms)
* Isolated stenosis of the anterior cerebral artery, posterior cerebral artery, MCA division, or a distal branch of the MCA
* Intracranial or extracranial arterial dissection, Moya Moya disease, vasculitis, radiation induced vasculopathy, fibromuscular dysplasia
* Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, dilated cardiomyopathy, left atrial spontaneous echo contrast
* A contraindication to the use of either warfarin or aspirin e.g. active peptic ulcer disease, active bleeding diathesis, platelets < 100,000*, hematocrit < 30*, clotting factor abnormality that increases the risk of bleeding, alcohol or substance abuse, severe gait instability, cerebral hemorrhage, systemic hemorrhage within the past year, severe liver impairment (SGOT > 3x normal*, cirrhosis), allergy to aspirin or warfarin, uncontrolled severe hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 115mm Hg), positive stool guaiac that is not attributable to hemorrhoids, creatinine > 3.0*
* Indication for intravenous heparin beyond randomization
* A severe neurological deficit that renders the patient incapable of living independently
* Dementia or psychiatric problem that prevents the patient from following an outpatient program reliably
* Co-morbid conditions that may limit survival to less than five years
* Pregnancy or female in age range of childbearing potential who is not using contraception
* Enrollment in another study that would conflict with the current study
* Excluded because difficult to measure percent stenosis of these small arteries, lesions are uncommon, and prognosis of patients - With these lesions is unknown * on most recent test done within 90 days prior to randomization, including day 90

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Marc Chimowitz, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States